CLINICAL TRIAL: NCT05517213
Title: High-dose Etoposide +G-CSF Versus High-dose Cyclophosphamide +G-CSF in Peripheral Blood Stem Cell Mobilization in Patients With Multiple Myeloma：a Multicenter,Randomized,Prospective Study
Brief Title: High-dose Chemotherapy+G-CSF in Peripheral Blood Stem Cell Mobilization in Patients With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 307-947168-89
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Etoposide; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: All patients were randomly assigned 1:1 to CTX 3.0g/m2+ G-CSF 10ug/kg or VP-16 1.2g/m2+G-CSF10ug/kg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Etoposide (Experimental): Etoposide1.2g/m2(Pump continuously for 24h)+G-CSF10ug/kg.
  Interventions: Drug: Etoposide
- Cyclophosphamide (Experimental): Cyclophosphamide 3.0g/m2+Grh-CSF10ug/kg.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Etoposide — Chemotherapy combined with rhG-CSF is widely used in autologous hematopoietic stem cell mobilization programs. For patients who do not meet the criteria of stem cell collection, they can be mobilized again after 1 month of rest. Chemotherapy +rhG-CSF mobilization or rhG-CSF+ ploxafo steady-state mobilization can be used.
  Other Names: VP-16
  Arms: Etoposide
Drug: Cyclophosphamide — Chemotherapy combined with rhG-CSF is widely used in autologous hematopoietic stem cell mobilization programs. For patients who do not meet the criteria of stem cell collection, they can be mobilized again after 1 month of rest. Chemotherapy +rhG-CSF mobilization or rhG-CSF+ ploxafo steady-state mobilization can be used.
  Other Names: CTX
  Arms: Cyclophosphamide

SUMMARY:
This study was a multi-center, randomized, prospective study. The purpose is to clarify that high-dose VP-16+G-CSF has better mobilization efficiency and less toxic and side effects compared with high-dose CTX+G-CSF, and minimize mobilization failure, so as to provide convenient and high-quality mobilization programs for clinical practice and enable more patients to enter the transplantation stage smoothly.

DETAILED DESCRIPTION:
Autologous peripheral blood hematopoietic stem cell mobilization: the two regiments were VP-16 1.2g/m2+rhG-CSF 10ug·kg-1·d-1 and CTX 3.0g/m2+rhG-CSF 10ug·kg-1·d-1; After high-dose chemotherapy, RHG-CSF 5ug/kg Bid was injected subcutaneously until the end of stem cell collection when the white blood cell count decreased to the minimum and began to rise steadily, and the platelet count was ≥50×109/L. Vp-16 was used as pure liquid continuously pumped for 24h. Dexamethasone 10mg was given before use, and blood pressure was monitored during use. During the use of CTX, it should be hydrated and alkalized, and mesic sodium (total amount 1.0-1.2 times CTX, divided into three static drops) should be used. Apheresis was performed once a day from the 5th day of RHG-CSF application, and the circulating blood volume was 2-3 times of the blood volume each time, and apheresis was performed at most 3 times. The percentage of CD34+ cells in the collection was determined by FCM, and the volume of the collection, the total number of nucleated cells per kg body weight and the number of CD34+ cells were recorded. For some patients whose apheresis is not up to the standard, they can be mobilized again after 1 month of rest, and chemotherapy +rhG-CSF mobilization or rhG-CSF+ ploxafo steady-state mobilization can be used.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MM patients: patients who were initially diagnosed and treated, who were suitable for autologous transplantation and planned to be treated with ASCT;

  * Age limitation: 18-70 years old patients; ④ Physical status: ECOG physical status score was 0 or 1; ⑤ The adverse reactions caused by chemotherapy had recovered: peripheral blood leukocytes ≥3.0×109/L, hemoglobin ≥80g/L, platelet ≥80×109/L; Liver function glutamic-pyruvic transaminase and glutamic-oxalacetic transaminase ≤ 2 times the upper limit of normal value, total bilirubin ≤ 1.5 times the upper limit of normal value, serum creatinine ≤ 1.5 times the upper limit of normal value, chest CT normal, ecg normal; (5) Patients participate voluntarily and informed consent is signed by patients themselves (or their legal representatives); Take effective contraceptive measures during the childbearing age.

Exclusion Criteria:

① According to the clinical judgment of the researcher: According to NCI CTCAE (4th edition May 28, 2009), patients with ≥3 grade cardiopulmonary insufficiency and severe kidney disease, currently diagnosed as coronary heart disease, myocardial infarction, arrhythmia, glutamic-oxalacetic transaminase, glutamic-pyruvic transaminase ≥ 2 times the upper limit of normal value, Total bilirubin ≥ 1.5 times the upper limit of normal;

* With active infection, including fever of unknown cause (axillary temperature > 37.5℃); ③ Patients with severe history of mental system.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Main purpose | Enrollment is expected to last for one year, followed up for two years.
  Compared with the literature data, The primary efficacy endpoint was the difference in the proportion of patients who reached the target CD34+ cells ≥5×106/kg and CD34+ cells ≥5×106/kg within 3 days of monotherapy between the study group and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital 307, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No